CLINICAL TRIAL: NCT05136833
Title: A Phase IIb Study to Explore the Efficacy and Safety of the Concomitant Administration of RUTI® Immunotherapy With the Standard Treatment in Patients With TB
Brief Title: Evaluation of Efficacy and Safety of the Concomitant of RUTI® Immunotherapy With the Standard Treatment in TB Patients
Acronym: CONSTAN
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Covid-19 pandemia
Sponsor: Archivel Farma S.L. (Industry)
Collaborators: Fundació Institut Germans Trias i Pujol (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-R6; 2021-003301-22 (EudraCT Number)
Record Dates: First submitted 2021-11-10; First posted 2021-11-29 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (RUTI) (Experimental): Subjets will receive one inoculation of the RUTI® vaccine at the same time as standard treatment is started. It will be administered subcutaneously in the deltoid region at a dose of 25 µg of fragmented, purified and liposomed heat-inactivated Mycobacterium tuberculosis bacilli (FCMtb) in an injection volume of 0.3 mL
  Interventions: Biological: RUTI® vaccine
- Group B (Placebo) (Placebo Comparator): Subjets will receive one inoculation of normal saline at the same time as standard treatment is started. It will be administered subcutaneously in the deltoid region.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: RUTI® vaccine — Each dose of the RUTI® vaccine contains 25 µg of fragmented, purified and liposomed heat-inactivated Mycobacterium tuberculosis bacilli (FCMtb) in a total volum of 0.3mL.
  Arms: Group A (RUTI)
Biological: Placebo — Normal saline will be used as a placebo.
  Arms: Group B (Placebo)

SUMMARY:
The study is an exploratory clinical trial to evaluate the efficacy and safety of the treatment with a vaccine against tuberculosis (RUTI®) given at the same time as standard treatment in patients with tuberculosis. It is a prospective, randomized (1:1), double-blind, multicentre, placebo-controlled clinical phase IIb trial.

DETAILED DESCRIPTION:
Patients will be randomized (1: 1) to receive an inoculation of RUTI® or placebo at the same time that standard treatment is started.

The standard TB treatment will continue after RUTI® or placebo administration according to SOC guidelines. All the patients will be followed up 6 months after the vaccination or until the end of SOC treatment.

Once all the patients have completed the week 2 follow-up, a Data Safety Monitoring Board (DSMB) will be established to review all relevant safety and toxicity data.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (females and males) aged ≥ 18.
2. Written informed consent in a language they understand. This includes informed consent to be in the trial and informed consent to collect specimens.
3. Laboratory confirmed pulmonary TB (with or without extrapulmonary involvement) defined as a hard copy of a sputum laboratory result that reports Mtb detection by sputum-microscopy smear-positive at least 1+, rapid molecular assay or mycobacterial culture.
4. Patients who have not received any anti-tubercular treatment in the last 24 hours.
5. Females of non-childbearing potential: at least 2 years post-menopausal or surgically sterile (e.g. tubal ligation).
6. Females of childbearing potential (including females less than 2 years post-menopausal) must have a negative pregnancy test at enrolment and must agree to use highly effective methods of birth control (i.e. diaphragm plus spermicide or male condom plus spermicide, oral contraceptive in combination with a second method, contraceptive implant, injectable contraceptive, indwelling intrauterine device, sexual abstinence, or a vasectomized partner) while participating in the study.
7. Males must agree to use a double-barrier method of contraception (condom plus spermicide or diaphragm plus spermicide) at least 1 month after RUTI/placebo vaccination; or the male patient or his female partner must be surgically sterile (e.g. vasectomy, tubal ligation) or the female partner must be post-menopausal.
8. The patient must be willing and able to attend all study visits and comply with all study procedures.

Exclusion Criteria:

1. Unable to provide written informed consent.
2. Women reported, or detected, or willing to be pregnant during the trial period.
3. Severity of illness precluding full evaluation: expected early death, evidenced by respiratory failure, low blood pressure, WHO performance score 3-4.
4. Bodyweight < 40kg.
5. Evidence of rifampicin resistance via GeneXpert.
6. Unstable Diabetes Mellitus as a poor metabolic control within the past 12 months.
7. For HIV infected subjects if the CD4+ count <250 cells/μL.
8. Major co-morbid conditions or any other finding which in the opinion of the investigator would compromise the protocol compliance or significantly influence the interpretation of results (i.e. cancer, immunodeficiency of any nature including treatment with immunosuppressant drugs and excluding HIV infection).
9. Any of the following laboratory parameters:

   * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 x upper limit of normal (ULN);
   * Total bilirubin > 2 x ULN;
   * Neutrophil count ≤ 500 neutrophils / mm3;
   * Platelet count < 50,000 platelets / mm3.
10. Alcohol use: potential participant either self-reports or in the investigator's opinion that the patient drinks more than an average of four units/day over a usual week or is a binge drinker (men: 5 or more drinks; women: consume 4 or more drinks, in about 2 hours).
11. Documented allergy to TB vaccines or any of the study treatment excipients, notably, to the RUTI® vaccine.
12. Concurrent enrolment in another clinical study, unless it is an observational (noninterventional) clinical study or during the follow-up period of an interventional study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Early Bactericidal Activity (EBA) from day 0 to day 14 | Daily between day 0 and day 14 after treatment initiation and RUTI®/placebo vaccination.
  Measured as the reduction of bacillary load of M. Tuberculosis based upon Time to detection (TTD) signal in MGIT.

SECONDARY OUTCOMES:
Early Bactericidal Activity (EBA) from 2 to 14 days | Daily between day 2 and day 14 after treatment initiation and RUTI®/placebo vaccination.
  Measured as the reduction of bacillary load of M. Tuberculosis based upon Time to detection (TTD) signal in MGIT. Difference between each intervention arm and control group.
Early Bactericidal Activity (EBA) from 7 to 14 days | Daily between day 7 and day 14 after treatment initiation and RUTI®/placebo vaccination.
  Measured as the reduction of the bacillary load of M. Tuberculosis based upon Time to detection (TTD) signal in MGIT.
Early Bactericidal Activity (EBA) from 4 to 24 week | At week 4, 8, 16 and 24 after treatment initiation and RUTI®/placebo vaccination
  Measured as the reduction of the bacillary load of M. Tuberculosis based upon Time to detection (TTD) signal in MGIT
Hazard ratio for stable culture conversion (SCC). | 24 weeks of TB treatment
  Difference between each intervention arm and control group.
Rate of Change in Time to Sputum Culture Positivity (TTP) in Liquid Culture Media (Days 0-14). | 14 days
  Difference between each intervention arm and control group.
Rate of Change in Time to Sputum Culture Positivity (TTP) in Liquid Culture Media (week 4, 8, 16 and 24 ) | Up to week 24
  Difference between each intervention arm and control group.
The proportion of patients with AEs between each intervention arm and the control group. | Up to week 24
  Difference of patients with AEs between each intervention arm and control group.
The proportion of patients with SAEs between each intervention arm and the control group | Up to week 24
  Difference of patients with SAEs between each intervention arm and control group.
Proportion of patients with CLINICAL, X-ray or LABORATORY worsening | Through study completion, an average of 24 weeks
  Difference of patients with Clinical, X-ray or Laboratory worsening between each intervention arm and control group.
Proportion of patients with improvement of clinical signs and symptoms, Bandim TB score | At weeks 2, 8, 24
  Difference of patients with improvement of clinical signs and symptoms between intervention and control group.
Number of patients with improvement of Health-related Quality of Life (HRQoL) comparing baseline measure with that over the course of therapy. | At week 8, week 24
  Difference f patients with improvement of HRQoL between each intervention arm and control group.

OTHER OUTCOMES:
IFN-γ production of ex vivo stimulated peripheral blood mononuclear cells (PBMC) (Exploratory endpoint for immunogenicity outcomes 1) | Up to week 24
  Immunogenic properties of the intervention group will be compared to the control group assessed by the evaluation of IFN-γ production of specific immune cells.
The summative ability of PBMCs to control mycobacterial growth inhibition assay (MGIA) (Exploratory endpoint for immunogenicity outcomes 2) | Up to week 24
  Immunogenic properties of the intervention group will be compared to the control group assessed by the summative ability of specific immune cells to control mycobacterial growth inhibition.